CLINICAL TRIAL: NCT01052753
Title: The Association Between Executive Functions and Candidate Genes of Dopaminergic and Noradrenergic Systems in Attention-deficit Hyperactivity Disorder
Brief Title: The Association Between Executive Functions and Candidate Genes of Dopaminergic and Noradrenergic Systems in Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 200912118R
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; executive function; endophenotype; dopaminergic system; noradrenergic system; candidate gene; Family-based association study
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD group
- Control group

SUMMARY:
The ultimate goal of this study is to find specific polymorphism of candidate genes (particularly of dopaminergic and noradrenergic systems) associated with intermediate phenotypes (e.g., executive functions, IQ, and other neuropsychological function) and/or phenomenological phenotypes (subtypes, comorbidity, dimensional approach) of ADHD. We propose to replicate the analysis of the candidate genes identified by previous genetic studies and recent findings from GWAS on ADHD using the candidate gene association study design (family-based case control study using parental controls and population-based case-control study). These results may lead our research team: (1) to resolve controversies over inconsistent findings in previous genetic studies and contribute to the literature on the validity of ADHD and its subtypes using clinical and genetic data; (2) to identify potential endophenotypes for ADHD genetic studies; and (3) to identify specific polymorphism of candidate genes and gene expressions of dopaminergic and noradrenergic systems associated with executive functions measured by the CANTAB.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a common, impairing, highly heritable, clinically heterogeneous early-onset neuropsychiatric disorder. Despite substantial evidence supporting genetic etiology of ADHD, molecular genetic studies so far have not yet provided any conclusive results using the categorical or subgroup approach of phenotype. Hence, there has been growing interest in using endophenotypes in molecular genetic studies on ADHD. Our previous studies have demonstrated significant deficits in executive functions among children with ADHD and the efficacy of methylphenidate and atomoxetine, involving dopaminergic and noradrenergic systems, in reducing ADHD core symptoms and improving executive functions. In a longitudinal follow-up family study on ADHD, we also reported that executive dysfunctions measured by the Cambridge Neuropsychological Test Automated Batteries (CANTAB) are potential endophenotypes for ADHD. Hence, identifying specific polymorphism of candidate genes of dopaminergic and noradrenergic systems associated with executive dysfunctions in Han Chinese in Taiwan is warranted.

Specific Aims:

1. To identify specific genetic polymorphism of candidate genes of dopaminergic and noradrenergic systems (e.g., DRD2, DRD4, DRD5, DAT1, NET, ADRA2A, DBH, COMT etc.) associated with executive dysfunctions measured by the CANTAB and other alternative phenotype approaches (ADHD subtypes, comorbidities, treatment effects, IQ, symptom dimensions and severity);
2. to investigate the relationship between a variety of ADHD phenotypes and endophenotypes and gene expressions of DRD2, DAT1, NET, ADRA2A, DBH, and COMT;
3. to validate executive functions and to search for other neuropsychological functioning as endophenotypes for ADHD; and
4. to determine whether ADHD is familial and identify which core symptoms of ADHD and which component of neuropsychological functioning are most familial;

Subjects and Methods: The major study design is the family-based case-control candidate gene association study. We will recruit 150 probands with ADHD, aged 7-18, and their parents (n = 300) and siblings (n= 150) and 150 school controls in three years (50, 60, and 40 families with ADHD and 50, 60, 40 school controls in the 1st, 2nd, and 3rd year, respectively). The measures include (1) interviews for psychopathology (K-SADS-E) and social functioning (SAICA), (2) self-administered questionnaires to measures ADHD symptoms (CPRS-R:S, CTRS-R:S, SNAP-IV and Adult ADHD rating scale) and comorbid conditions (ASRI and CBCL), and (3) neuropsychological tests: WISC-III-R, CPT, CANTAB, and Time Perception Tasks. The transmission/disequilibrium test (TDT) and quantitative TDT by using FBAT and FBAT-GEE, GEE, and Mixed Models will be used for data analysis.

Anticipated Results: We anticipate the establishment of clinical, neuropsychological, and genetic database of at least 350 families (150 families in this project) and 150 same-age controls, the completion of genetic analysis and gene expressions of several candidate genes including those involving dopaminergic and noradrenergic systems, and identification of genetic variants for ADHD diagnosis, symptoms, and comorbidities, executive functions, and other neurocognitive endophenotypes in a Taiwanese sample. The findings of different approaches to identify the genetic etiologies for ADHD in this study should help us determine the most promising approach for future molecular genetic studies on ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the proband subjects are (1) that subjects have a clinical diagnosis of ADHD, or Hyperkinetic Disorder (HD) defined by the DSM-IV and ICD-10, respectively, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits; (2) their ages range from 7 to 18 when we conduct the study; (3) subjects who are able to perform the CANAB and time tests; (4) subjects' IQ greater than 80; (5) subjects have both biological parents; (6) both parents are Han Chinese; and (7) subjects and their biological parents (and siblings if any) consent to participate in this study for complete phenotype assessments and blood data collection.
* The inclusion criteria for the control subjects are (1) that subjects who do not have the diagnosis of ADHD, or Hyperkinetic Disorder (HD) defined by the DSM-IV and ICD-10, respectively, in the past and current assessments; (2) subjects who are able to perform the CANAB and time tests; (4) subjects' IQ greater than 80; (5) subjects are Han Chinese; and (6) subjects and their mothers consent to participate in this study for complete phenotype assessments.

Exclusion Criteria:

* The proband subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, or Pervasive Developmental Disorder. Moreover, the subjects will also be excluded from the study if they completely cannot cooperate with blood withdrawal or neuropsychological assessments.
* The control subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, or Pervasive Developmental Disorder. Moreover, the subjects will also be excluded from the study if they completely cannot cooperate with neuropsychological assessments.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The proband sample will consist of at least 150 drug-naïve children and adolescents with ADHD, aged 7-18 (who are able to perform the CANTAB and time tasks) from Department of Psychiatry, National Taiwan University Hospital (NTUH). Their biological parents (n = 300) and siblings (estimated number = 150) born to the same biological parents will be recruited as the parent controls and sibling controls, respectively, for the family-based case control study. We will recruit 150 school controls without lifetime diagnosis of ADHD in the same school districts and with similar age and gender distributions of the probands with ADHD.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan